CLINICAL TRIAL: NCT03637257
Title: Measurement of Expired Carbon Dioxide: Comparison of a Modified CO2/O2 Guedel Airway With a Nasal Cannula in Sedated Children Aged 4-24 Months
Brief Title: Carbon Dioxide (CO2) Measurement With a CO2/O2 Guedel Airway
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to other priorities
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UKBB_Anae_CO2_Gued_Feas
Record Dates: First submitted 2018-08-07; First posted 2018-08-17 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Breathing Stop
Keywords: Capnography; Pediatric; nasal cannula; Guedel airway
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blinded cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal cannula / Guedel (Experimental): Record of capnography using a standard nasal cannula followed by use of a modified Guedel airway
  Interventions: Device: modified Guedel airway
- Guedel / nasal cannula (Experimental): Record of capnography using a modified Guedel airway followed by use of a standard nasal cannula
  Interventions: Device: modified Guedel airway

INTERVENTIONS:
Device: modified Guedel airway — Monitoring of breathing

SUMMARY:
This trial compares capnographic signals using a modified CO2/O2 Guedel airway with a CO2/O2 nasal cannula without and with oxygen supply in sedated children aged 4 - 24 months.

DETAILED DESCRIPTION:
Sedation of pediatric patients is frequently jeopardized by respiratory adverse events such as central and/or obstructive apnea resulting in hypoxemia. Various factors such as patient comorbidities, medication and inconsistent physiologic monitoring are known to contribute to or facilitate adverse events during sedation. Therefore, monitoring of breathing by capnography is recommended and has become common standard e.g. by the use of a CO2/O2 nasal cannula.

However, capnography derived from CO2/O2 nasal cannulas may be impaired and these impairments are exaggerated in infants based on their physiologic characteristics (small tidal volumes, high respiratory rates).

To overcome these impairments, the investigators developed a modified CO2/O2 Guedel airway including a CO2 sampling port at the tip of the airway. In a previous study, significantly more accurate capnographic signals resulted compared with measurements derived from a nasal cannula when using a modified CO2/O2 Guedel airway in a model of a breathing 6-month-old manikin.

The aim of the study is to examine the accuracy of capnographic measurements of the modified CO2/O2 Guedel airway in comparison with measurements from a CO2/O2 nasal cannula in sedated children aged 4 - 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Term born infants aged 4 to 24 months
* Physical status according classification I or II (American Society of Anaesthesiologists (ASA))
* Scheduled for elective diagnostic/therapeutic procedures or surgery under sedation/anaesthesia
* Informed Consent as documented by signature of the parents or legal caregiver

Exclusion Criteria:

* syndrome that affects the airway anatomy
* Physical status according classification III or IV (American Society of Anaesthesiologists (ASA))
* Upper respiratory tract infection at present or within the last two weeks before the study
* Previous enrolment into the current study
* Known hypersensitivity or allergic reactions to midazolam, nitrous oxide (N2O), Propofol or Sevoflurane.
* Positive Family History for malignant hyperthermia, Morbus Pompe or ophthalmic operations with gas injection or Sinus- or inner ear surgery.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
end-tidal carbon-dioxide concentration (etCO2) | 90 seconds
  Difference between capillary and maximum etCO2 sampled via a modified CO2/O2 Guedel airway versus a CO2/O2 nasal cannula

SECONDARY OUTCOMES:
Change of end-tidal carbon-dioxide concentration (etCO2) according to different oxygen flows (O2) | 90 seconds
  Effect of O2 administration on etCO2 measurement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Erb, Prof. Dr. MD, Principal Investigator — UKBB
Locations (1):
- University Children´s Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll J, Anagnostopoulou P, Frei FJ, Erb TO. A modified CO2/O2 Guedel airway improves capnographic accuracy compared with a CO2/O2 nasal cannula: An infant manikin study. Eur J Anaesthesiol. 2018 Aug;35(8):566-572. doi: 10.1097/EJA.0000000000000818. PMID 29757925